CLINICAL TRIAL: NCT05453383
Title: Clinical Recruitment of Patients With First-line Targeted Drug Resistance or Intolerance to Hepatocellular Cancer With PD-1 Inhibitor (Toripalimab,JS001) Detected on the NGS Platform Combined With Anlotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shen Feng (Other)
Responsible Party: Sponsor-Investigator, Shen Feng, Director of Oncology Department, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-201908
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Cancer
Keywords: Antotinib Toripalimab
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib and Toripalimab treatment (Experimental): Anlotinib Hydrochloride and Toripalimab Injection
  Interventions: Drug: Anlotinib;Toripalimab

INTERVENTIONS:
Drug: Anlotinib;Toripalimab — Anlotinib Hydrochloride;Toripalimab injiection
  Other Names: AL3818;JS001

SUMMARY:
PD-1 inhibitors have become the standard treatment for advanced hepatocellular cancer, while targeted drugs such as sorafenib and lenvatinib are the first-line standard treatment for hepatocellular cancer. Recent studies have shown that PD-1 inhibitors combined with targeted drugs can improve the efficacy of hepatocellular cancer.To clear the joint treatment in patients with advanced hepatocellular cancer (HCC) efficacy and evaluate its safety, we proposed to carry out the PD - 1 inhibitor (Toripalimab, JS001) joint anti-angiogenesis small molecules targeting drug anlotinib for clinical research,at the same time, based on joint solution of NGS platform testing to predict the curative effect, bring benefit for the long-term survival of patients with hepatocellular cancer (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of hepatocellular cancer;
2. At least one measurable lesion was assessed according to RECIST1.1 criteria.
3. Age from 18 to 75,ECOG physical strength score reaches 0-2;
4. After first-line targeted therapy, it was assessed as advanced or intolerant according to RECIST1.1 criteria.
5. Child-pugh grade A or B for liver function;
6. Bone marrow function was basically normal: neutrophils > 1.5x 10^9/L, platelets > 75 x10^9/L;
7. Adequate renal reserve: creatinine <130 mol/L;
8. Centerless dysfunction, chest pain (medically uncontrollable), no myocardial infarction within 12 months prior to study initiation;
9. Estimated survival ≥3 months;
10. Signed the informed consent.

Exclusion Criteria:

1. Previous application of PD-1 inhibitor and anlotinib;
2. Secondary malignant tumors or other tumors (except superficial skin cancer and localized low-grade malignant tumors) occurring within 3 years prior to the start of the study;
3. Metastasis of the brain or meninges;
4. Imaging findings indicated that the tumor was involved in important blood vessels or that the researchers had assessed that it might lead to fatal bleeding during follow-up;
5. Bleeding events at any site ≥CTCAE level 3 occurred 4 weeks before medication, and there were unhealed wounds, ulcers or fractures;
6. The time of occurrence of arteriovenous thrombosis, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism, within 6 months before enrollment;
7. Untreated intestinal obstruction or subobstruction that cannot eat or affect systemic administration;
8. Patients with active infection or other possible disorders receive inflammatory infections under planned management;
9. Have a history of uncontrolled substance abuse or mental disorders;
10. In the judgment of the investigator, patients with concomitant diseases that may seriously endanger their own safety or may affect the completion of the study;
11. Participated in other clinical trials;
12. Pregnant and nursing women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-08 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | at least 2 months
  Objective response rate include response from stable disease to complete

SECONDARY OUTCOMES:
Progression-free survival | at least 2 months
  The time between the start of randomization and tumorigenesis or death

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China